CLINICAL TRIAL: NCT01055041
Title: A Randomized, Open Labeled Comparative Study to Assess the Efficacy and Safety of Controller Medications as Add on to Inhaled Steroid and Long Acting β2 Agonist in Treatment of Moderate to Severe Persistent Bronchial Asthma
Brief Title: Controller Medications in the Management of Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Bhavnagar (Other)
Responsible Party: Dr. C. B. Tripathi, Professor and Head , Department of Pharmacology, Government Medical College, Bhavnagar-364001, Gujarat, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pharmacol no.03 /2008 Research
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Moderate to Severe Persistent Bronchial Asthma
MeSH Terms: interventions — montelukast; doxofylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- inhaled budesonide and formeterol plus oral montelukast (Experimental): 1st two weeks -run in period .All three participants prescribed Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day Next 8 weeks- Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day plus tablet montelukast (10 mg/day)orally in the evening
  Interventions: Drug: inhaled budesonide and formeterol plus oral montelukast
- inhaled budesonide and formeterol plus oral doxophylline (Experimental): 1st two weeks -run in period, all three participants prescribed Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day Next 8 weeks
  Interventions: Drug: inhaled budesonide and formeterol plus oral doxophylline
- Doubling the dose of inhaled budesonide and formeterol (Experimental): 1st two weeks -run in period all the participants prescribed Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day Next 8 weeks- Metered dose inhaler (budesonide 200 mcg /puff + formeterol 6 mcg/puff) two times a day plus metered dose inhaler of budesonide (200 mcg/puff) two times a day
  Interventions: Drug: Doubling the dose of inhaled budesonide and formeterol

INTERVENTIONS:
Drug: inhaled budesonide and formeterol plus oral montelukast — 1st two weeks -run in period all the participants prescribed Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day Next 8 weeks- Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day plus tablet montelukast (10 mg/day)orally in the evening
  Arms: inhaled budesonide and formeterol plus oral montelukast
Drug: inhaled budesonide and formeterol plus oral doxophylline — 1st two weeks -run in period, all participants prescribed Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day Next 8 weeks- Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day plus tablet doxophylline sustained release(400 mg/day)orally in the morning
  Arms: inhaled budesonide and formeterol plus oral doxophylline
Drug: Doubling the dose of inhaled budesonide and formeterol — 1st two weeks -run in period, all groups participants prescribed Metered dose inhaler (budesonide 200 mcg/puff + formeterol 6 mcg/puff) two times a day Next 8 weeks- Metered dose inhaler (budesonide 200 mcg /puff + formeterol 6 mcg/puff) two times a day plus metered dose inhaler of budesonide (200 mcg/puff) two times a day
  Arms: Doubling the dose of inhaled budesonide and formeterol

SUMMARY:
The purpose of this study is to know the effect of another controller medication add on to the inhaled corticosteroid and long acting β2 agonist on clinical symptom, lung function and compliance in patients of moderate to severe persistent bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

* aged between 15 to 65 years of either sex
* had clinically diagnosed Bronchial asthma
* had poor asthma control defined by ACQ score (asthma control questionnaire) of 1.5 or greater
* FEV1 (Forced Expiratory Volume at 1 second) value of 50% or more of predicted
* improvement in FEV1 was greater than 15% after bronchodilator inhalation

Exclusion Criteria:

* major illness of system other than respiratory major respiratory illness other than asthma taken long acting anti histaminic within a preceding week of enrollment Smokers Pregnant and lactating woman history of hypersensitivity to any of above drugs

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome was percentage of improvement in FEV1 | 10 weeks

SECONDARY OUTCOMES:
Improvement in PEFR (Peak expiratory flow rate), ACQ scores(asthma control questionnaire score), rates of adverse drug reaction and EPACs (episodes of poor asthma control) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yogesh A Patel, M.B.B.S, Principal Investigator — Sir T. General Hospital and Government Medical College, Bhavnagar-364001, Gujarat, India; Dr. Chandrabhanu R Tripathi, MD, Study Chair — Professor and Head, Department of Pharmacology, Government Medical College, Bhavnagar-364001, Gujarat, India
Locations (1):
- Sir Takthasinhji General Hospital Bhavnagar, Gujarat, India, Bhavnagar, Gujarat, India